CLINICAL TRIAL: NCT04245787
Title: Remineralization Potential of Curodont Repair Flouride Plus Versus CPP-ACP in Management of White Spot Lesions: Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Hamada Ahmed Shehab Eldin, resident at operative dentistry department, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p11 4
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: White Spot Lesion
MeSH Terms: interventions — Fluorides

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self assembling peptide with fluoride (Experimental)
  Interventions: Drug: Self assembling peptide with fluoride
- Casein-phosphopeptide/amorphous-calcium phosphate (Active Comparator)
  Interventions: Drug: Self assembling peptide with fluoride

INTERVENTIONS:
Drug: Self assembling peptide with fluoride — peptide forms a 3D matrix within demineralized carious lesions areas, which enables novo hydroxyapatite crystal formation facilitating the so-called guided enamel regeneration of the lost enamel structure. The peptide has shown encouraging results as a scaffold for enamel regeneration
  Other Names: Curodont Repair Fluoride Plus

SUMMARY:
The goal of modern dentistry is to manage non-cavitated caries lesions non- invasively through re-mineralization process to prevent the disease progression and improve aesthetics, strength, and function. Re-mineralization is defined as the process that supplies calcium, phosphate and flouride ions from an external source to the tooth to convert ion deposition into crystal voids in demineralized enamel. White spot lesions should be managed using a multifactorial approach. The most important strategy is to prevent demineralization and biofilm formationand use of methodologies for remineralization of lesions .

Self-assembling peptide (P11-4) has shown great potential for natural repair of early caries lesions through emerging biomimetic re-mineralization properties. (Takahashi Fet al in 2015) This peptide forms a 3D matrix within demineralized carious lesions areas, which enables novo hydroxyapatite crystal formation facilitating the so-called guided enamel regeneration of the lost enamel structure. The peptide has shown encouraging results as a scaffold for enamel regeneration

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35 years of age female and males
* Had received conventional periodontal therapy
* Active carious white spot lesions
* No systemic diseases or concomitant medication affecting salivary flow

Exclusion Criteria:

* - Participant in another trial
* Non carious lesion (enamel hypoplasia and dental flourosis)
* Presence of abnormal oral, medical, or mental condition.
* Participants who had evidence of reduced salivary flow or significant tooth wear.
* Allergy to MI paste

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Remineralization potential | T0:baseline assessment -->T1:1 month (Assessment of white spot lesion regression)--> T2:4 months(Application of Curodont repair flouride plus /Cpp-Acp andAssessment of white spot lesion regression)--> T3: 6 months Assessment of white spot lesion regres(
  by: Inspection under magnification ICDAS II Score 0:Sound tooth surface:
  1. First visual change in enamel.
  2. Distinct visual change in enamel visible when wet, lesion must be visible when dry.

SECONDARY OUTCOMES:
Remineralization potential | T0:baseline assessment -->T1:1 month (Assessment of white spot lesion regression)--> T2:4 months(Application of Curodont repair flouride plus /Cpp-Acp andAssessment of white spot lesion regression)--> T3: 6 months( Assessment of white spot lesion regres
  by: Image analysis software Change in area of the white spot lesion (mm2)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Oral & Dental Medicine - Cairo University, Cairo, Egypt